CLINICAL TRIAL: NCT01900977
Title: Population Effects of Antiretroviral Therapy to Reduce HIV Transmission (PopART): A Cluster-randomized Trial of the Impact of a Combination Prevention Package on Population-level HIV Incidence in Zambia and South Africa
Brief Title: Population Effects of Antiretroviral Therapy to Reduce HIV Transmission (PopART)
Acronym: PopART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HIV Prevention Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Drug Abuse (NIDA) (NIH); Office of the U.S. Global AIDS Coordinator (Unknown); Bill and Melinda Gates Foundation (Other); London School of Hygiene and Tropical Medicine (Other); Imperial College London (Other); Zambart (Other); Desmond Tutu TB Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 071; 11865 (Other: DAIDS-ES); UM1AI068619 (NIH)
Record Dates: First submitted 2013-07-02; First posted 2013-07-17 (Estimated); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: HIV
Keywords: Universal Test and Treat (UTT); Combination Prevention
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A Universal Testing w/Immediate ART (Active Comparator)
  Interventions: Other: Universal Testing with immediate ART
- Arm B ART according to National Guidelines (Active Comparator)
  Interventions: Other: Universal Testing with ART eligibility according to National Guidelines
- Standard of Care (Other): Includes:
  Strengthening of HIV testing and ART services according to national guidelines at health facilities and other venues; Strengthening of male circumcision and PMTCT services available at health facilities and other venues in the community; and Treatment of STIs and provision of condoms at health facilities and other venues in the community.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Universal Testing with immediate ART — • Combination prevention package including:
  o House-to-house deployment of: Universal HIV counseling and testing; Active linkage to care for individuals diagnosed as HIV-infected, with immediate eligibility for ART; Promotion of male circumcision and prevention of mother to child transmission (PMTCT) services; Provision of condoms; Strengthening of HIV testing and services at health facilities and other venues; Strengthening of male circumcision and prevention of mother-to-child transmission of HIV services available in the community; and Treatment of sexually transmitted infections (STIs) and provision of condoms at health units
  Other Names: PopART Intervention; UTT
  Arms: Arm A Universal Testing w/Immediate ART
Other: Universal Testing with ART eligibility according to National Guidelines — Combination prevention package including:
  House-to-house deployment of: Universal HIV counseling and testing; Active linkage to care for individuals diagnosed as HIV-infected, with ART eligibility according to national guidelines; Promotion of male circumcision and PMTCT services; Provision of condoms; Strengthening of HIV testing and services at health facilities and other venues; Strengthening of male circumcision and PMTCT services available in the community; and Treatment of STIs and provision of condoms at health units.
  Other Names: PopART Intervention
  Arms: Arm B ART according to National Guidelines
Other: Standard of Care
  Arms: Standard of Care

SUMMARY:
PopART is a community randomized trial that is investigating whether a community-wide combination HIV prevention package including annual home-based HIV testing, active referral and the offer of immediate ART for those testing HIV-positive, along with the promotion of proven HIV prevention methods (such as voluntary medical male circumcision, prevention of mother to child transmission and condom use), will help to prevent transmission and substantially reduce new HIV infections. The study is being conducted in 21 communities in Zambia and South Africa (randomized into 3 arms, each with 7 communities) with a total population of approximately 1.2 million individuals.

DETAILED DESCRIPTION:
HIV Prevention Trials Network (HPTN) 071 (PopART) will investigate the impact on HIV incidence of universal voluntary HIV counseling and testing (with referral to care) provided to a community through a house-to-house campaign, in combination with early ART for individuals who are HIV-positive, and other proven preventive interventions. The design of HPTN 071 (PopART) will allow the study team to distinguish between the impact of universal testing with referral for HIV care in accordance with national guidelines, and the impact of universal testing with referral for early ART initiation for those with HIV infection. In addition, HPTN 071 (PopART) will determine if a program of universal voluntary testing, including early ART initiation, is feasible and acceptable when delivered on a large scale to entire communities. Evaluating the effectiveness of universal voluntary HIV counseling and testing with the offer of early ART is a key global health priority.

ELIGIBILITY:
Inclusion Criteria:

1. Population Cohort

   1. 18 - 44 years of age
   2. Able and willing to provide informed consent
   3. Residing within catchment area of a designated local health unit and intending to remain so for the next three years
   4. Residing in a randomly selected household
2. Case-Control Study 1 Inclusion Criteria:

   1. At least 18 years of age
   2. Able and willing to provide informed consent
   3. Resident in the cluster during the first round of testing
   4. Visited by a CHiP team and offered testing during the first round of home-based testing
3. Case-Control Study 2 Inclusion Criteria:

   1. At least 18 years of age
   2. Able and willing to provide informed consent
   3. Resident in the cluster during the first round of testing
   4. Tested HIV-infected in CHiP home-based testing, or HIV-infected and disclosed that they were previously diagnosed as HIV-infected to CHiP team
4. Case-Control Study 3 Inclusion Criteria:

   1. At least 18 years of age
   2. Able and willing to provide informed consent
   3. Resident in the cluster during the second round of testing
   4. Visited by a CHiP team and offered testing during the second round of home-based testing

Exclusion Criteria:

1. Population Cohort Exclusion Criteria:

   1. Current or planned enrollment in another HIV treatment, prevention, or Pre-Exposure Prophylaxis (PrEP) study
   2. Current, planned or prior enrollment in an HIV vaccine study
   3. Anything that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
2. Case-Control Study 1 Exclusion Criteria:

   1. Individuals belonging to the Population Cohort or other case-control studies
   2. Individuals known to be HIV-infected after testing elsewhere.
3. Case-Control Study 2 Exclusion Criteria:

   1. Individuals enrolled in the Population Cohort or other case-control studies
   2. HIV-infected individuals already on ART before study commences
4. Case-Control Study 3 Exclusion Criteria:

   1. Known HIV infected from CHiP data.
   2. Individuals belonging to the Population Cohort or other case-control studies

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48540 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-07-07 (Actual); Study Completion 2018-07-07 (Actual)

PRIMARY OUTCOMES:
HIV incidence measured over 3 years in the Population Cohort, with the primary analysis including HIV incidence measured between Months 12 and 36 of the study. | 3 years

SECONDARY OUTCOMES:
HIV incidence over the first, second, and third years of follow-up | 3 years
ART adherence and viral suppression | 24 months
  HIV viral load at 24 months in HIV-infected members of the Population Cohort who initiated HIV care and ART after commencement of the PopART intervention in the community (if funding available)
Herpes Simplex Virus -2 (HSV-2) incidence | 12 months, 24 months, and 36 months
  Incident HSV-2 infections at 12 months, 24 months, and 36 months for all individuals in the Population Cohort who were HSV-2-uninfected at enrollment
HIV disease progression, retention in care, and death | 3 years
ART toxicity | 3 years
  ART safety and clinical events among Population Cohort participants initiating ART after commencement of the PopART intervention in the community, measured using routine health center data, and
  ART safety and clinical events among health center attendees who initiated ART after commencement of the PopART intervention in the community, measured using routine health center data
Sexual risk behavior | 3 years
  o Self-reported sexual risk behavior at Enrollment, 12 months, 24 months, and 36 months in the Population Cohort
Case notification rate of tuberculosis (TB) | 3 years
  * Case notification rates of bacteriologically-confirmed TB diagnosed among the general population of patients seeking care at health centers as recorded by health centers
  * TB mortality among TB cases in the community as recorded by health centers
HIV-related stigma | 3 years
  * Self-reported data on stigma indicators at enrollment, 12 months, 24 months, and 36 months in the Population Cohort
  * Qualitative interviews in selected members of the general population in Arms A, B, and
Uptake of PMTCT | 3 years
  * Self-reported use of services for PMTCT at Enrollment, 12 months, 24 months, and 36 months among HIV-infected women in the Population Cohort who had been pregnant in the prior 12 months
  * Uptake of PMTCT services at health centers
  * Uptake of PMTCT as indicated in data collected in households by CHiPs
Uptake of male circumcision | 3 years
  * Self-reported circumcision status/uptake at Enrollment, 12 months, 24 months, and 36 months of men in the Population Cohort
  * Uptake of circumcision in the community as indicated in health center data
  * Uptake of circumcision as indicated in data collected in households by CHiPs
ART screening and uptake | 3 years
  * The proportion of Population Cohort members, identified as HIV-infected who screen for ART eligibility, and who subsequently initiate ART
  * Proportion of community members, identified as HIV-infected in data from CHiP teams, who screen for ART eligibility, and who subsequently initiate ART, as indicated in health center data
HIV testing and retesting | 3 years
  * Self-reported recent HIV testing at Enrollment, 12 months, 24 months, and 36 months in the Population Cohort
  * The number of adults (16 years and older) in the household and the number of HIV tests performed as indicated in data from CHiP teams and health centers
Time between HIV diagnosis and initiation of care | 3 years
  * The proportion of Population Cohort members initiating HIV care within 3 months of a positive HIV diagnosis
  * The proportion of community members initiating HIV care within 3 months of HIV diagnosis as indicated in data from CHiP teams (provision of HIV positive result) and health center data (date of care initiation)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hayes, BSc, MSc, DSc, Study Chair — London School of Hygiene and Tropical Medicine; Sarah Fidler, MBBS, PhD, Study Chair — Imperial College London; Helen Ayles, BSc, MBBS, MSc, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Nulda Beyers, MBChB, FCP, MSc, PhD, Principal Investigator — Stellenbosch Univeristy; Peter Bock, MD, MRCP, MRCGP, MPH, PhD, Principal Investigator — University of Stellenbosch
Locations (2):
- Desmund Tutu TB Centre at Stellenbosch University, Cape Town, Western Cape, South Africa
- Zambart, Lusaka, Zambia

REFERENCES:
- [Background] Bond V, Hoddinott G, Viljoen L, Simuyaba M, Musheke M, Seeley J. Good Health and Moral Responsibility: Key Concepts Underlying the Interpretation of Treatment as Prevention in South Africa and Zambia Before Rolling Out Universal HIV Testing and Treatment. AIDS Patient Care STDS. 2016 Sep;30(9):425-34. doi: 10.1089/apc.2016.0114. PMID 27610464
- [Background] Hargreaves JR, Stangl A, Bond V, Hoddinott G, Krishnaratne S, Mathema H, Moyo M, Viljoen L, Brady L, Sievwright K, Horn L, Sabapathy K, Ayles H, Beyers N, Bock P, Fidler S, Griffith S, Seeley J, Hayes R; HPTN 071 (PopART) study team. HIV-related stigma and universal testing and treatment for HIV prevention and care: design of an implementation science evaluation nested in the HPTN 071 (PopART) cluster-randomized trial in Zambia and South Africa. Health Policy Plan. 2016 Dec;31(10):1342-1354. doi: 10.1093/heapol/czw071. Epub 2016 Jul 3. PMID 27375126
- [Background] Viljoen L, Thorne M, Thomas A, Bond V, Hoddinott G; HPTN 071 (PopART) team. A narrative analysis positioning HIV relative to personal (sexual) relationship challenges in an agony aunt column in the Western Cape, South Africa - Aunty Mona's "love advice". AIDS Care. 2016;28 Suppl 3:83-9. doi: 10.1080/09540121.2016.1178957. PMID 27421055
- [Background] Camlin CS, Seeley J, Viljoen L, Vernooij E, Simwinga M, Reynolds L, Reis R, Plank R, Orne-Gliemann J, McGrath N, Larmarange J, Hoddinott G, Getahun M, Charlebois ED, Bond V. Strengthening universal HIV 'test-and-treat' approaches with social science research. AIDS. 2016 Mar 27;30(6):969-70. doi: 10.1097/QAD.0000000000001008. No abstract available. PMID 26959355
- [Background] Hayes R, Ayles H, Beyers N, Sabapathy K, Floyd S, Shanaube K, Bock P, Griffith S, Moore A, Watson-Jones D, Fraser C, Vermund SH, Fidler S; HPTN 071 (PopART) Study Team. HPTN 071 (PopART): rationale and design of a cluster-randomised trial of the population impact of an HIV combination prevention intervention including universal testing and treatment - a study protocol for a cluster randomised trial. Trials. 2014 Feb 13;15:57. doi: 10.1186/1745-6215-15-57. PMID 24524229
- [Background] Cori A, Ayles H, Beyers N, Schaap A, Floyd S, Sabapathy K, Eaton JW, Hauck K, Smith P, Griffith S, Moore A, Donnell D, Vermund SH, Fidler S, Hayes R, Fraser C; HPTN 071 PopART Study Team. HPTN 071 (PopART): a cluster-randomized trial of the population impact of an HIV combination prevention intervention including universal testing and treatment: mathematical model. PLoS One. 2014 Jan 15;9(1):e84511. doi: 10.1371/journal.pone.0084511. eCollection 2014. PMID 24454728
- [Background] Vermund SH, Fidler SJ, Ayles H, Beyers N, Hayes RJ. Can combination prevention strategies reduce HIV transmission in generalized epidemic settings in Africa? The HPTN 071 (PopART) study plan in South Africa and Zambia. J Acquir Immune Defic Syndr. 2013 Jul;63 Suppl 2(0 2):S221-7. doi: 10.1097/QAI.0b013e318299c3f4. PMID 23764639
- [Background] Vermund SH, Hayes RJ. Combination prevention: new hope for stopping the epidemic. Curr HIV/AIDS Rep. 2013 Jun;10(2):169-86. doi: 10.1007/s11904-013-0155-y. PMID 23456730
- [Background] Sabapathy K, Van den Bergh R, Fidler S, Hayes R, Ford N. Uptake of home-based voluntary HIV testing in sub-Saharan Africa: a systematic review and meta-analysis. PLoS Med. 2012;9(12):e1001351. doi: 10.1371/journal.pmed.1001351. Epub 2012 Dec 4. PMID 23226107
- [Background] Hayes R, Sabapathy K, Fidler S. Universal testing and treatment as an HIV prevention strategy: research questions and methods. Curr HIV Res. 2011 Sep;9(6):429-45. doi: 10.2174/157016211798038515. PMID 21999778
- [Result] Hoddinott G, Myburgh H, de Villiers L, Ndubani R, Mantantana J, Thomas A, Mbewe M, Ayles H, Bock P, Seeley J, Shanaube K, Hargreaves J, Bond V, Reynolds L; HPTN 071 (PopART) Study Team. Households, fluidity, and HIV service delivery in Zambia and South Africa - an exploratory analysis of longitudinal qualitative data from the HPTN 071 (PopART) trial. J Int AIDS Soc. 2018 Jul;21 Suppl 4(Suppl Suppl 4):e25135. doi: 10.1002/jia2.25135. PMID 30027687
- [Result] Bond V, Ngwenya F, Thomas A, Simuyaba M, Hoddinott G, Fidler S, Hayes R, Ayles H, Seeley J; HPTN 071 (PopART) study team. Spinning plates: livelihood mobility, household responsibility and anti-retroviral treatment in an urban Zambian community during the HPTN 071 (PopART) study. J Int AIDS Soc. 2018 Jul;21 Suppl 4(Suppl Suppl 4):e25117. doi: 10.1002/jia2.25117. PMID 30027643
- [Result] Floyd S, Ayles H, Schaap A, Shanaube K, MacLeod D, Phiri M, Griffith S, Bock P, Beyers N, Fidler S, Hayes R; HPTN 071 (PopART) Study Team. Towards 90-90: Findings after two years of the HPTN 071 (PopART) cluster-randomized trial of a universal testing-and-treatment intervention in Zambia. PLoS One. 2018 Aug 10;13(8):e0197904. doi: 10.1371/journal.pone.0197904. eCollection 2018. PMID 30096139
- [Result] Sabapathy K, Mulubwa C, Mathema H, Mubekapi-Musadaidzwa C, Schaap A, Hoddinott G, Hargreaves J, Floyd S, Ayles H, Hayes R; HPTN 071 (PopART) Study Team. Is home-based HIV testing universally acceptable? Findings from a case-control study nested within the HPTN 071 (PopART) trial. Trop Med Int Health. 2018 Jun;23(6):678-690. doi: 10.1111/tmi.13055. Epub 2018 Apr 16. PMID 29608231
- [Result] Bock P, Fatti G, Ford N, Jennings K, Kruger J, Gunst C, Louis F, Grobbelaar N, Shanaube K, Floyd S, Grimwood A, Hayes R, Ayles H, Fidler S, Beyers N; HPTN 071 (PopART) trial team. Attrition when providing antiretroviral treatment at CD4 counts >500cells/muL at three government clinics included in the HPTN 071 (PopART) trial in South Africa. PLoS One. 2018 Apr 19;13(4):e0195127. doi: 10.1371/journal.pone.0195127. eCollection 2018. PMID 29672542
- [Result] Bradley J, Floyd S, Piwowar-Manning E, Laeyendecker O, Young A, Bell-Mandla N, Bwalya J, Bock P, Fidler S, Ayles H, Hayes RJ; HPTN 071 (PopART) Study Team. Sexually Transmitted Bedfellows: Exquisite Association Between HIV and Herpes Simplex Virus Type 2 in 21 Communities in Southern Africa in the HIV Prevention Trials Network 071 (PopART) Study. J Infect Dis. 2018 Jul 2;218(3):443-452. doi: 10.1093/infdis/jiy178. PMID 29659909
- [Result] Hargreaves JR, Krishnaratne S, Mathema H, Lilleston PS, Sievwright K, Mandla N, Mainga T, Vermaak R, Piwowar-Manning E, Schaap A, Donnell D, Ayles H, Hayes RJ, Hoddinott G, Bond V, Stangl A; HPTN 071 (PopART) Study Team. Individual and community-level risk factors for HIV stigma in 21 Zambian and South African communities: analysis of data from the HPTN071 (PopART) study. AIDS. 2018 Mar 27;32(6):783-793. doi: 10.1097/QAD.0000000000001757. PMID 29369164
- [Result] Bock P, Jennings K, Vermaak R, Cox H, Meintjes G, Fatti G, Kruger J, De Azevedo V, Maschilla L, Louis F, Gunst C, Grobbelaar N, Dunbar R, Limbada M, Floyd S, Grimwood A, Ayles H, Hayes R, Fidler S, Beyers N. Incidence of Tuberculosis Among HIV-Positive Individuals Initiating Antiretroviral Treatment at Higher CD4 Counts in the HPTN 071 (PopART) Trial in South Africa. J Acquir Immune Defic Syndr. 2018 Jan 1;77(1):93-101. doi: 10.1097/QAI.0000000000001560. PMID 29016524
- [Result] Viljoen L, Ndubani R, Bond V, Seeley J, Reynolds L, Hoddinott G. Community narratives about women and HIV risk in 21 high-burden communities in Zambia and South Africa. Int J Womens Health. 2017 Nov 29;9:861-870. doi: 10.2147/IJWH.S143397. eCollection 2017. PMID 29238230
- [Result] Sabapathy K, Mubekapi-Musadaidzwa C, Mulubwa C, Schaap A, Hoddinott G, Stangl A, Floyd S, Ayles H, Fidler S, Hayes R; HPTN 071 (PopART) study team. Predictors of timely linkage-to-ART within universal test and treat in the HPTN 071 (PopART) trial in Zambia and South Africa: findings from a nested case-control study. J Int AIDS Soc. 2017 Dec;20(4):e25037. doi: 10.1002/jia2.25037. PMID 29251433
- [Result] Thomas R, Burger R, Harper A, Kanema S, Mwenge L, Vanqa N, Bell-Mandla N, Smith PC, Floyd S, Bock P, Ayles H, Beyers N, Donnell D, Fidler S, Hayes R, Hauck K; HPTN 071 (PopART) Study Team. Differences in health-related quality of life between HIV-positive and HIV-negative people in Zambia and South Africa: a cross-sectional baseline survey of the HPTN 071 (PopART) trial. Lancet Glob Health. 2017 Nov;5(11):e1133-e1141. doi: 10.1016/S2214-109X(17)30367-4. Epub 2017 Sep 27. PMID 28964756
- [Result] Bock P, Phiri C, Piwowar-Manning E, Kosloff B, Mandla N, Young A, James A, Schaap A, Scheepers M, Donnell D, Griffith S, El-Sadr W, Shanaube K, Beyers N, Hayes R, Fidler S, Ayles H; HPTN 071 (PopART) Study Team. Understanding low sensitivity of community-based HIV rapid testing: experiences from the HPTN 071 (PopART) trial in Zambia and South Africa. J Int AIDS Soc. 2017 Aug 29;20(Suppl 6):21780. doi: 10.7448/IAS.20.7.21780. PMID 28872272
- [Result] Shanaube K, Schaap A, Chaila MJ, Floyd S, Mackworth-Young C, Hoddinott G, Hayes R, Fidler S, Ayles H; HPTN 071 (PopART) Study Team. Community intervention improves knowledge of HIV status of adolescents in Zambia: findings from HPTN 071-PopART for youth study. AIDS. 2017 Jul 1;31 Suppl 3(Suppl 3):S221-S232. doi: 10.1097/QAD.0000000000001530. PMID 28665880
- [Result] Shanaube K, Schaap A, Floyd S, Phiri M, Griffith S, Chaila J, Bock P, Hayes R, Fidler S, Ayles H; HPTN 071 (PopART) Study Team. What works - reaching universal HIV testing: lessons from HPTN 071 (PopART) trial in Zambia. AIDS. 2017 Jul 17;31(11):1555-1564. doi: 10.1097/QAD.0000000000001514. PMID 28471766
- [Result] Hayes R, Floyd S, Schaap A, Shanaube K, Bock P, Sabapathy K, Griffith S, Donnell D, Piwowar-Manning E, El-Sadr W, Beyers N, Ayles H, Fidler S; HPTN 071 (PopART) Study Team. A universal testing and treatment intervention to improve HIV control: One-year results from intervention communities in Zambia in the HPTN 071 (PopART) cluster-randomised trial. PLoS Med. 2017 May 2;14(5):e1002292. doi: 10.1371/journal.pmed.1002292. eCollection 2017 May. PMID 28464041
- [Result] Simwinga M, Bond V, Makola N, Hoddinott G, Belemu S, White R, Shanaube K, Seeley J, Moore A; HPTN 071 (PopART) study team. Implementing Community Engagement for Combination Prevention: Lessons Learnt From the First Year of the HPTN 071 (PopART) Community-Randomized Study. Curr HIV/AIDS Rep. 2016 Aug;13(4):194-201. doi: 10.1007/s11904-016-0322-z. PMID 27405816
- [Result] Bond V, Chiti B, Hoddinott G, Reynolds L, Schaap A, Simuyaba M, Ndubani R, Viljoen L, Simwinga M, Fidler S, Hayes R, Ayles H, Seeley J; HPTN 071 (PopART) study team. "The difference that makes a difference": highlighting the role of variable contexts within an HIV Prevention Community Randomised Trial (HPTN 071/PopART) in 21 study communities in Zambia and South Africa. AIDS Care. 2016;28 Suppl 3:99-107. doi: 10.1080/09540121.2016.1178958. PMID 27421057
- [Derived] Burger R, Bell-Mandla N, Harper A, Richardson S, Kanema S, Thomas R, Mwenge L, Wilson E, Floyd S, Bock P, Ayles H, Fidler S, Hayes R, Hauck K; HPTN 071 (PopART) study team. Does enhanced HIV prevention, diagnosis, and linkage to care reduce hospitalisation in high HIV-burden communities in Zambia and South Africa? findings from the HPTN 071 (PopART) randomised trial. PLOS Glob Public Health. 2025 May 8;5(5):e0004373. doi: 10.1371/journal.pgph.0004373. eCollection 2025. PMID 40339051
- [Derived] Skalland TM, de Dieu Tapsoba J, Zangeneh SZ, Floyd S, Ayles H, Bock P, Fidler S, Eshleman SH, Hayes RJ, Donnell D; HPTN 071 (PopART) Study Team. A survey weighted analysis of HPTN 071 (PopART) primary outcome of HIV incidence. AIDS Res Ther. 2025 Mar 7;22(1):30. doi: 10.1186/s12981-025-00720-0. PMID 40055795
- [Derived] Steinhaus MC, Nicholson TJ, Pliakas T, Harper A, Lilleston P, Mainga T, Milimo D, Jennings K, Grobbelaar N, Louis F, Liebenberg H, Hayes RJ, Fidler S, Ayles H, Bock P, Hoddinott G, Hargreaves JR, Bond V, Stangl AL; HPTN 071 (PopART) study team. Prevalence and risk of burnout among HIV service providers in South Africa and Zambia: findings from the HPTN 071 (PopART) trial. Hum Resour Health. 2024 Jul 8;22(1):50. doi: 10.1186/s12960-024-00934-9. PMID 38978065
- [Derived] Telisinghe L, Floyd S, MacLeod D, Schaap A, Dunbar R, Bwalya J, Bell-Mandla N, Piwowar-Manning E, Donnell D, Shaunaube K, Bock P, Fidler S, Hayes RJ, Ayles HM; HPTN 071 (PopART) study team. Incidence of self-reported tuberculosis treatment with community-wide universal testing and treatment for HIV and tuberculosis screening in Zambia and South Africa: A planned analysis of the HPTN 071 (PopART) cluster-randomised trial. PLoS Med. 2024 May 31;21(5):e1004393. doi: 10.1371/journal.pmed.1004393. eCollection 2024 May. PMID 38820246
- [Derived] Chaila MJ, Mcleod D, Vermund SH, Mbolongwe-Thornicroft M, Mbewe M, Mubekapi-Musadaidzwa C, Harper A, Schaap A, Floyd S, Hoddinott G, Hayes R, Fidler S, Ayles H, Shanaube K; HPTN 071 (PopART) for Youth (P-ART-Y) Study Team. Assessment of a screening tool to aid home-based identification of adolescents (aged 10-14) living with HIV in Zambia and South Africa: HPTN 071 (PopART) study. PLoS One. 2024 Feb 16;19(2):e0266573. doi: 10.1371/journal.pone.0266573. eCollection 2024. PMID 38363733
- [Derived] Klinkenberg E, Floyd S, Shanaube K, Mureithi L, Gachie T, de Haas P, Kosloff B, Dodd PJ, Ruperez M, Wapamesa C, Burnett JM, Kalisvaart N, Kasese N, Vermaak R, Schaap A, Fidler S, Hayes R, Ayles H; TREATS study team. Tuberculosis prevalence after 4 years of population-wide systematic TB symptom screening and universal testing and treatment for HIV in the HPTN 071 (PopART) community-randomised trial in Zambia and South Africa: A cross-sectional survey (TREATS). PLoS Med. 2023 Sep 8;20(9):e1004278. doi: 10.1371/journal.pmed.1004278. eCollection 2023 Sep. PMID 37682971
- [Derived] Skalland T, Ayles H, Bock P, Bwalya J, Shanaube K, Kasese N, Dupre M, Kosloff B, Floyd S, Wilson E, Moore A, Eshleman S, Fidler S, Hayes R, Donnell D; HPTN 071 (PopART) Study Team. Community- and individual-level correlates of HIV incidence in HPTN 071 (PopART). J Int AIDS Soc. 2023 Aug;26(8):e26155. doi: 10.1002/jia2.26155. PMID 37643290
- [Derived] Yang B, Sloot R, Floyd S, Awoniyi D, Griffith S, Ayles H, Fidler S, Hayes R, Vermund SH, Bock P; HPTN 071 (PopART) study team. Brief Report: How Do We Reach Men? Offering HIV Testing in Evenings and Weekends in the HPTN 071 (PopART) Community-Based Trial in South Africa. J Acquir Immune Defic Syndr. 2023 Aug 1;93(4):300-304. doi: 10.1097/QAI.0000000000003197. PMID 37001128
- [Derived] Wilson E, Donnell D, Skalland T, Floyd S, Moore A, Bell-Mandla N, Bwalya J, Kasese N, Dunbar R, Shanaube K, Kosloff B, Laeyendecker O, Agyei Y, Hoddinott G, Bock P, Fidler S, Hayes R, Ayles H; HPTN 071 (PopART) Study Team. Impact of universal testing and treatment on sexual risk behaviour and herpes simplex virus type 2: a prespecified secondary outcomes analysis of the HPTN 071 (PopART) community-randomised trial. Lancet HIV. 2022 Nov;9(11):e760-e770. doi: 10.1016/S2352-3018(22)00253-3. PMID 36332653
- [Derived] Donnell D. Practical issues in operationalizing the design and outcome evaluation of cluster randomized trials. Clin Trials. 2022 Aug;19(4):407-415. doi: 10.1177/17407745221087465. Epub 2022 Apr 8. PMID 35393864
- [Derived] Phiri MM, Schaap A, Simwinga M, Hensen B, Floyd S, Mulubwa C, Simuyaba M, Chiti B, Bond V, Shanaube K, Fidler S, Hayes R, Ayles H; HPTN 071 (PopART) Study team. Closing the gap: did delivery approaches complementary to home-based testing reach men with HIV testing services during and after the HPTN 071 (PopART) trial in Zambia? J Int AIDS Soc. 2022 Jan;25(1):e25855. doi: 10.1002/jia2.25855. PMID 35001530
- [Derived] Bell-Mandla NF, Sloot R, Maarman G, Griffith S, Moore A, Floyd S, Hayes R, Fidler S, Ayles H, Bock P; HPTN 071 (PopART) study team. Improving retention of community-recruited participants in HIV prevention research through Saturday household visits; findings from the HPTN 071 (PopART) study in South Africa. BMC Med Res Methodol. 2021 Nov 8;21(1):242. doi: 10.1186/s12874-021-01415-6. PMID 34749654
- [Derived] Bond V, Hoddinott G, Viljoen L, Ngwenya F, Simuyaba M, Chiti B, Ndubani R, Makola N, Donnell D, Schaap A, Floyd S, Hargreaves J, Shanaube K, Fidler S, Bock P, Ayles H, Hayes R, Simwinga M, Seeley J; HPTN071 (PopART) study team. How 'place' matters for addressing the HIV epidemic: evidence from the HPTN 071 (PopART) cluster-randomised controlled trial in Zambia and South Africa. Trials. 2021 Apr 6;22(1):251. doi: 10.1186/s13063-021-05198-5. PMID 33823907
- [Derived] Stangl AL, Pliakas T, Mainga T, Steinhaus M, Mubekapi-Musadaidzwa C, Viljoen L, Dunbar R, Schaap A, Floyd S, Mandla N, Bond V, Hoddinott G, Fidler S, Hayes R, Ayles H, Bock P, Donnell D, Hargreaves JR; HPTN 071 (PopART) study team. The effect of universal testing and treatment on HIV stigma in 21 communities in Zambia and South Africa. AIDS. 2020 Nov 15;34(14):2125-2135. doi: 10.1097/QAD.0000000000002658. PMID 32773484
- [Derived] Jones HS, Floyd S, Stangl A, Bond V, Hoddinott G, Pliakas T, Bwalya J, Mandla N, Moore A, Donnell D, Bock P, Fidler S, Hayes R, Ayles H, Hargreaves JR; HPTN 071 (PopART) Study Team. Association between HIV stigma and antiretroviral therapy adherence among adults living with HIV: baseline findings from the HPTN 071 (PopART) trial in Zambia and South Africa. Trop Med Int Health. 2020 Oct;25(10):1246-1260. doi: 10.1111/tmi.13473. Epub 2020 Aug 26. PMID 32745296
- [Derived] Floyd S, Shanaube K, Yang B, Schaap A, Griffith S, Phiri M, Macleod D, Sloot R, Sabapathy K, Bond V, Bock P, Ayles H, Fidler S, Hayes R; HPTN 071 (PopART) study team. HIV testing and treatment coverage achieved after 4 years across 14 urban and peri-urban communities in Zambia and South Africa: An analysis of findings from the HPTN 071 (PopART) trial. PLoS Med. 2020 Apr 2;17(4):e1003067. doi: 10.1371/journal.pmed.1003067. eCollection 2020 Apr. PMID 32240156
- [Derived] Eshleman SH, Piwowar-Manning E, Wilson EA, Lennon D, Fogel JM, Agyei Y, Sullivan PA, Weng L, Moore A, Laeyendecker O, Kosloff B, Bwalya J, Maarman G, van Deventer A, Floyd S, Bock P, Ayles H, Fidler S, Hayes R, Donnell D; HPTN 071 (PopART) Study Team. Determination of HIV status and identification of incident HIV infections in a large, community-randomized trial: HPTN 071 (PopART). J Int AIDS Soc. 2020 Feb;23(2):e25452. doi: 10.1002/jia2.25452. PMID 32072743
- [Derived] Stangl AL, Lilleston P, Mathema H, Pliakas T, Krishnaratne S, Sievwright K, Bell-Mandla N, Vermaak R, Mainga T, Steinhaus M, Donnell D, Schaap A, Bock P, Ayles H, Hayes R, Hoddinott G, Bond V, Hargreaves JR; HPTN 071 (PopART) Study Team. Development of parallel measures to assess HIV stigma and discrimination among people living with HIV, community members and health workers in the HPTN 071 (PopART) trial in Zambia and South Africa. J Int AIDS Soc. 2019 Dec;22(12):e25421. doi: 10.1002/jia2.25421. PMID 31840400
- [Derived] Hayes RJ, Donnell D, Floyd S, Mandla N, Bwalya J, Sabapathy K, Yang B, Phiri M, Schaap A, Eshleman SH, Piwowar-Manning E, Kosloff B, James A, Skalland T, Wilson E, Emel L, Macleod D, Dunbar R, Simwinga M, Makola N, Bond V, Hoddinott G, Moore A, Griffith S, Deshmane Sista N, Vermund SH, El-Sadr W, Burns DN, Hargreaves JR, Hauck K, Fraser C, Shanaube K, Bock P, Beyers N, Ayles H, Fidler S; HPTN 071 (PopART) Study Team. Effect of Universal Testing and Treatment on HIV Incidence - HPTN 071 (PopART). N Engl J Med. 2019 Jul 18;381(3):207-218. doi: 10.1056/NEJMoa1814556. PMID 31314965
- [Derived] Fatti G, Grimwood A, Nachega JB, Nelson JA, LaSorda K, van Zyl G, Grobbelaar N, Ayles H, Hayes R, Beyers N, Fidler S, Bock P. Better Virological Outcomes Among People Living With Human Immunodeficiency Virus (HIV) Initiating Early Antiretroviral Treatment (CD4 Counts >/=500 Cells/microL) in the HIV Prevention Trials Network 071 (PopART) Trial in South Africa. Clin Infect Dis. 2020 Jan 16;70(3):395-403. doi: 10.1093/cid/ciz214. PMID 30877753

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2015-11-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT01900977/Prot_ICF_000.pdf